CLINICAL TRIAL: NCT02195856
Title: The Effect of Dietary Nitrate on Hepatic Perfusion and Incretin Secretion
Brief Title: Effects of Nitrate on Liver Perfusion and Sugar Control
Acronym: DiMPLe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: Royal Devon and Exeter NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: CRF163; 14/SW/0092 (Other: NIHR Exeter Clinical Research Facility)
Record Dates: First submitted 2014-06-27; First posted 2014-07-21 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Type 2 Diabetes; Ageing
Keywords: Diabetes; Nitrate; Nitrite; Hepatic; MRI; Incretin; Insulin; Glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diseased condition (Active Comparator): Crossover design where participants will start in the Beetroot juice condition, and after a washout period, move into the other condition.
  Interventions: Dietary Supplement: Beetroot juice
- Placebo (Placebo Comparator): Crossover design where participants will start in the placebo condition, and after a washout period, move into the other condition.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Beetroot juice — 140mL concentrated Beetroot juice or placebo juice
  Other Names: James Whites Drinks Ltd
  Arms: Diseased condition
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Rationale:

Mediterranean style diets and diets rich in green leafy vegetables protect against the risk of developing type 2 diabetes and a wide range of cardiovascular disease. These diets are rich in nitrate. Numerous studies have shown that nitrate from the diet can have a wide range of beneficial effects. These include relaxing blood vessels and improving their function. It has been shown that following a meal with added nitrate, blood flow to the stomach increases more than would be expected if the same meal is given without nitrate. This is because when we eat nitrate the body concentrates it and recycles it through the digestive system. As it cycles through it is converted into nitrite and nitric oxide which cause blood vessels to relax. The nitrite and nitric oxide also seem to protect against infection from food sources such as E.coli.

What we do not know is whether this nitrite and nitric oxide has any effect on the small intestine and the liver. Some nitrite reaches the small intestine and may have the same effect on blood flow there as it does in the stomach. This could be very important because the small intestine releases hormones called incretins which we now know play a very important role in controlling blood sugar every time we eat. These incretin hormones regulate insulin release and the body's sensitivity to insulin. When we eat blood containing the substances we have absorbed from the gut, such as sugars and fats, goes to the liver for processing. The blood then leaves the liver and enters the circulation. This means the blood supply to the liver will have much higher concentrations of nitrite than the blood circulating in the rest of the body. High concentrations of nitrite appear to cause blood vessels to open up. This means more blood vessels in the liver should be opened after a nitrate rich meal. It seems likely that this will help the liver to control blood sugar more effectively.

Purpose To find out if supplementation by inorganic nitrate as found in beetroot or green leafy vegetables increases liver (hepatic) microvascular perfusion and increases incretin secretion.

Plan of investigations:

We will recruit 16 individuals for each of the three groups (Young adults, older adults and individuals with type 2 diabetes). Participants will be recruited from a database of volunteers who have consented to being contacted for research studies which are held by the NIHR Exeter Clinical Research Facility. This is a double blind, placebo controlled crossover design study (nitrate rich beetroot juice vs a placebo, nitrate depleted beetroot juice). Three visits will be required for participants to complete this study.

Visit 1. Screening and consent. The experimenter will explain to the participant what the study is designed to test. If the participant is completely clear on the study and understand what they are agreeing to, they will sign a consent form. In addition a standard medical history and clinical examination will be undertaken by a research nurse and or Anthony Shepherd. A venous blood sample will be taken using standard aseptic procedures. Following consent participants will be assigned a study number. Study numbers will be previously assigned (by a research statistician) to a randomisation order to begin either the beetroot juice or placebo arm of the study first.

Visit 2. Visit 2 will require the participant to fast over night from 10pm. Only water will be admissible from this time. The following morning participants will arrive at the laboratory in a fully hydrated and rested state at ~ 7.30am. This visit will take ~ 5 hours and will require 4 MRI scans. Participants will have the first MRI scan after a short acclimatisation period. Participants will then be provided with a concentrated 140 mL nitrate drink or placebo with a standardised breakfast (2 slices of toast with butter). Three subsequent MRI scans will be required (one per hour for three hours). Venous blood samples taken from cannulas will be sampled, in order to assess glucose, insulin, incretins and nitrate/nitrite prior to each scan. Visit 3. Visit 3 will take place after a minimum washout period of 7 days from Visit 2. Visit 3 will be identical in nature to visit 2; however, it will be with the opposite supplement (either nitrate rich or placebo beetroot juice).

Impact:

Dietary nitrate appears to offer a simple, low cost means of modifying cardiovascular risk. This study will deepen our understanding of the role of the nitrate/nitrite/nitric oxide pathway in normal physiology. By understanding what effect inorganic nitrate from the diet has on hepatic perfusion and other pathways involved in glucose homeostasis this may lead to a range of simple, low cost therapeutic strategies to prevent and treat type 2 diabetes.

DETAILED DESCRIPTION:
Hypothesis

Inorganic nitrate from the diet, following conversion to nitrite and nitric oxide via the pathways described above will:

1. Increase hepatic microvascular perfusion
2. Increase GLP-1 secretion
3. Increase pancreatic insulin secretion
4. Reduce the area under the curve for glucose post meal

Purpose To find out if inorganic nitrate found in green leafy vegetables protect against the risk of developing type 2 diabetes and cardiovascular disease by increasing hepatic microvascular perfusion and increasing incretin secretion.

Aim The purpose of this study is to see if inorganic nitrate from the diet modulates hepatic perfusion and other pathways involved in post-prandial glucose homeostasis.

MRI Hepatic micro vessel perfusion of the liver and portal vein diameter will be measured by Dr. Jon Fulford at the Peninsula Magnetic Resonance Research Centre, St Luke's Campus. Following initial survey images to obtain anatomical information apparent diffusion coefficients (ADC) are calculated in the posterior right lobe of the liver. Diffusion images are acquired with a single shot echo-planar imaging (EPI) sequence with 15 directions and b values of 200 and 800 s mm-2. Images are acquired during a single breathe-hold at an axial-oblique orientation with a repetition time (TR) of 1500 ms an echo time of 57 ms, an in-plane resolution of 4 x 4 mm and a slice thickness of 10 mm with fat suppression and 3 signal averages.

ADC is given by:

ADC = 1/(b200-b800) Ln (S800/S200) where S800 is the signal with a diffusion b-value of 800 s mm-2 (b800) and S200 is the signal with a diffusion b-value of 200 s mm-2 (b200).

Statistical analysis Statistical analysis will be performed by an experienced and trained researcher and statistical advice will be available from Prof. Angela Shore from within the team and Beverly Shields from the NIHR Exeter Clinical Research Facility. Data will be assessed for normality. Depending on the normality of data the differences between the groups will be assessed by either unpaired t-test or Mann-Whitney test.

Sample Size Sixteen participants would need to be recruited per group in order to detect a 1SD difference between groups data with 80% power and an a of 0.05. Twenty participants would be recruited in order to account for drop outs.

ELIGIBILITY:
Inclusion Criteria:

* 1. Type 2 Diabetes group; aged between 35 - 75. Able to give informed consent 2. Older adults group; aged between 50 - 75. Not on any regular vasoactive medication and able to give informed consent. 3. Young adults group; aged between18 - 35. Not on any regular vasoactive medication and able to give informed consent.

Exclusion Criteria:

* • Antibiotic therapy within the preceding two weeks

  * Anyone on GLP-1 analogues or DPP4 inhibitors
  * Myocardial infarction or cerebro-vascular event within the preceding three months
  * Current smoker (any smoking event in last 3 months)
  * Previous brain surgery, cardiac pacemaker.
  * Metal fragments in the eye from previous injury
  * Severe claustrophobia
  * Uncontrolled hypertension
  * On regular organic nitrates, thiazolidinidiones or nicorandil
  * eGFR < 30
  * Any other serious medical condition which would interfere with data interpretation or safety.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-07; Primary Completion 2015-03-09 (Actual); Study Completion 2017-07-20 (Actual)

PRIMARY OUTCOMES:
Hepatic perfusion | 12 minutes
  Each participant will have 2 visits to the MRI facility. On each visit, they will have 4 scans lasting 12 minutes each.

SECONDARY OUTCOMES:
Plasma glucose concentration | 2 minutes
  Each participant will have 2 visits to the MRI facility. On each visit, they will have 4 scans lasting 12 minutes each. Just before each scan, venous blood samples will be drawn to assess plasma glucose concentration.
Plasma insulin concentration | 2 minutes
  Each participant will have 2 visits to the MRI facility. On each visit, they will have 4 scans lasting 12 minutes each. Just before each scan, venous blood samples will be drawn to assess plasma insulin concentration
Plasma incretin concentration | 2 minutes
  Each participant will have 2 visits to the MRI facility. On each visit, they will have 4 scans lasting 12 minutes each. Just before each scan, venous blood samples will be drawn to assess plasma incretin concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Angela C Shore, PhD, Study Chair — University of Exeter; Anthony I Shepherd, MSc, Principal Investigator — University of Exeter
Locations (2):
- United Kingdom (2):
  - Exeter Magnetic Resonance Research Centre, St Luke's Campus, Exeter, Devon
  - NIHR Exeter Clinical Research Facility, Exeter, Devon